CLINICAL TRIAL: NCT04623775
Title: A Phase 2 Randomized Study of Relatlimab Plus Nivolumab in Combination With Chemotherapy vs. Nivolumab in Combination With Chemotherapy as First Line Treatment for Participants With Stage IV or Recurrent Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Relatlimab Plus Nivolumab in Combination With Chemotherapy vs. Nivolumab in Combination With Chemotherapy as First Line Treatment for Participants With Stage IV or Recurrent Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA224-104; 2020-004026-31 (EudraCT Number); U1111-1256-8115 (Registry Identifier: WHO)
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer
Keywords: Stage IV Non-small Cell Lunch Cancer; Recurrent Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer; Relatlimab; Nivolumab; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; relatlimab; Carboplatin; Cisplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Arm A (Nivolumab + Relatlimab Dose 1 + Platinum Doublet Chemotherapy (PDCT)) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Pemetrexed
- Part 1: Arm B (Nivolumab + Relatlimab Dose 2 + PDCT)) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-Paclitaxel; Drug: Pemetrexed
- Part 2: Arm C (Nivolumab + Relatlimab Dose 2 + PDCT) (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed
- Part 2: Arm D (Nivolumab + PDCT) (Active Comparator)
  Interventions: Biological: Nivolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
Biological: Relatlimab — Specified dose on specified days
  Arms: Part 1: Arm A (Nivolumab + Relatlimab Dose 1 + Platinum Doublet Chemotherapy (PDCT)); Part 1: Arm B (Nivolumab + Relatlimab Dose 2 + PDCT)); Part 2: Arm C (Nivolumab + Relatlimab Dose 2 + PDCT)
Drug: Carboplatin — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
Drug: Cisplatin — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
Drug: Paclitaxel — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
Drug: Nab-Paclitaxel — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.
  Arms: Part 1: Arm A (Nivolumab + Relatlimab Dose 1 + Platinum Doublet Chemotherapy (PDCT)); Part 1: Arm B (Nivolumab + Relatlimab Dose 2 + PDCT))
Drug: Pemetrexed — Specified dose on specified days. Participant will receive only two of the listed chemotherapies (carboplatin, cisplatin, paclitaxel, nab-paclitaxel) along with immunotherapy.

SUMMARY:
The purpose of this study is to assess the safety profile of relatlimab plus nivolumab in combination with platinum doublet chemotherapy (PDCT) and to determine if nivolumab plus relatlimab in combination with PDCT improves overall response rate (ORR) when compared to nivolumab plus PDCT in participants with previously untreated Stage IV or recurrent non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed metastatic non-small cell lung cancer (NSCLC) of squamous (SQ) or non-squamous (NSQ) histology with Stage IV A/B (as defined by the 8th International Association for the Study of Lung Cancer Classification) or recurrent disease following multi-modal therapy for locally advanced disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of less than or equal to 1 at screening and confirmed prior to randomization.
* Measurable disease by computed tomography (CT) or magnetic resonance resources (MRI) per response evaluation criteria in solid tumor version 1.1 (RECIST 1.1) criteria.
* No prior systemic anti-cancer treatment (including epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) inhibitors) given as primary therapy for advanced or metastatic disease.

Exclusion Criteria

* Participants with EGFR, ALK, ROS-1, or known B-rapidly accelerated fibrosarcoma proto-oncogene (BRAF V600E) mutations that are sensitive to available targeted therapy.
* Untreated CNS metastases.
* Leptomeningeal metastases (carcinomatous meningitis).
* Concurrent malignancy requiring treatment or history of prior malignancy active within 2 years prior to randomization (ie, participants with a history of prior malignancy are eligible if treatment was completed at least 2 years before randomization and the participant has no evidence of disease).
* Prior treatment with an anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti-programmed death-ligand 2 (PD-L2), or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2026-02-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (125):
- United States (29):
  - Local Institution - 0160, Duarte, California
  - Local Institution - 0081, Orange, California
  - Local Institution - 0139, New Haven, Connecticut
  - Local Institution - 0153, Jacksonville, Florida
  - Local Institution - 0011, Port Saint Lucie, Florida
  - Local Institution - 0089, Athens, Georgia
  - Local Institution - 0121, Wichita, Kansas
  - Local Institution - 0159, Lexington, Kentucky
  - Local Institution - 0002, Louisville, Kentucky
  - Local Institution - 0082, Scarborough, Maine
  - Local Institution - 0129, Omaha, Nebraska
  - Local Institution - 0152, Howell Township, New Jersey
  - Local Institution - 0124, Johnson City, New York
  - Local Institution - 0162, Mineola, New York
  - Local Institution - 0128, New York, New York
  - Local Institution - 0165, New York, New York
  - Local Institution - 0097, The Bronx, New York
  - Local Institution - 0117, Durham, North Carolina
  - Local Institution - 0156, Cincinnati, Ohio
  - Local Institution - 0155, Cleveland, Ohio
  - Local Institution - 0084, Lancaster, Pennsylvania
  - Local Institution - 0147, Pittsburgh, Pennsylvania
  - Local Institution - 0148, Providence, Rhode Island
  - Local Institution - 0083, Greenville, South Carolina
  - Local Institution - 0149, Dallas, Texas
  - Local Institution - 0091, Harlingen, Texas
  - Local Institution - 0001, Tyler, Texas
  - Local Institution - 0092, Spokane, Washington
  - Local Institution - 0157, Morgantown, West Virginia
- Argentina (8):
  - Local Institution - 0037, Río Cuarto, Córdoba Province
  - Local Institution - 0021, Buenos Aires, Distrito Federal
  - Local Institution - 0014, Cuiudad Autonoma de Buenos Aires, Distrito Federal
  - Local Institution - 0039, Viedma, Río Negro Province
  - Local Institution - 0029, Rosario, Santa Fe Province
  - Local Institution - 0060, Córdoba
  - Local Institution - 0038, Córdoba
  - Local Institution - 0073, La Rioja
- Australia (10):
  - Local Institution - 0055, Camperdown, New South Wales
  - Local Institution - 0086, Gosford, New South Wales
  - Local Institution - 0132, Tamworth, New South Wales
  - Local Institution - 0057, Adelaide, South Australia
  - Local Institution - 0130, Ballarat, Victoria
  - Local Institution - 0138, Bendigo, Victoria
  - Local Institution - 0141, Box Hill, Victoria
  - Local Institution - 0109, Frankston, Victoria
  - Local Institution - 0119, Murdoch, Western Australia
  - Local Institution - 0085, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0090, Graz
  - Local Institution - 0126, Vienna
- Belgium (3):
  - Local Institution - 0127, Ghent
  - Local Institution - 0131, Ghent
  - Local Institution - 0125, Roeselare
- Brazil (9):
  - Local Institution - 0063, Natal, Rio Grande do Norte
  - Local Institution - 0161, Ijuí, Rio Grande do Sul
  - Local Institution - 0116, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0112, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0107, Barretos, São Paulo
  - Local Institution - 0111, Santo André, São Paulo
  - Local Institution - 0072, Rio de Janeiro
  - Local Institution - 0163, São Paulo
  - Local Institution - 0120, São Paulo
- Chile (3):
  - Local Institution - 0079, Santiago, Santiago Metropolitan
  - Local Institution - 0041, Santiago, Santiago Metropolitan
  - Local Institution - 0016, Santiago, Santiago Metropolitan
- France (7):
  - Local Institution - 0008, Rennes, Ille-Et-Vilaine
  - Local Institution - 0007, Dijon
  - Local Institution - 0144, Le Mans
  - Local Institution - 0102, Paris
  - Local Institution - 0035, Paris
  - Local Institution - 0006, Saint-Mandé
  - Local Institution - 0110, Paris, Île-de-France Region
- Germany (9):
  - Local Institution - 0065, Essen, North Rhine-Westphalia
  - Local Institution - 0103, Berlin
  - Local Institution - 0045, Berlin
  - Local Institution - 0062, Großhansdorf
  - Local Institution - 0058, Homburg
  - Local Institution - 0108, Löwenstein
  - Local Institution - 0071, Marburg
  - Local Institution - 0050, Paderborn
  - Local Institution - 0030, Ravensburg
- Ireland (2):
  - Local Institution - 0133, Elm Park, Dublin
  - Local Institution - 0023, Dublin
- Italy (7):
  - Local Institution - 0106, Rome, RA
  - Local Institution - 0028, Candiolo
  - Local Institution - 0009, Catania
  - Local Institution - 0032, Genova
  - Local Institution - 0059, Milan
  - Local Institution - 0164, Pesaro
  - Local Institution - 0019, Siena
- Mexico (4):
  - Local Institution - 0070, Mexico City, Mexico City
  - Local Institution - 0115, Monterrey, Nuevo León
  - Local Institution - 0013, San Pedro Garza García, Nuevo León
  - Local Institution - 0020, Toluca, State of Mexico
- Netherlands (2):
  - Local Institution - 0053, Harderwijk, Gelderland
  - Local Institution - 0158, Arnhem
- Poland (5):
  - Local Institution - 0145, Gdynia
  - Local Institution - 0036, Lublin
  - Local Institution - 0031, Lublin
  - Local Institution - 0080, Olsztyn
  - Local Institution - 0088, Warsaw
- Romania (5):
  - Local Institution - 0099, Cluj-Napoca, Cluj
  - Local Institution - 0017, Craiova, Dolj
  - Local Institution - 0012, Craiova, Jud. Dolj
  - Local Institution - 0069, Timișoara, Timiș County
  - Local Institution - 0052, Craiova
- Russia (3):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - LLC Eurocityclinic, Saint Petersburg
  - FSBI &quot,Research Institute of Influenza named after A.A. Smorodintsev &quot,of the MoH of the Rus, Saint Petersburg
- Spain (11):
  - Local Institution - 0075, Seville, Andalusia
  - Local Institution - 0137, Badalona, Barcelona
  - Local Institution - 0024, Barcelona, Catalonia
  - Local Institution - 0051, A Coruña
  - Local Institution - 0154, Barcelona
  - Local Institution - 0048, Barcelona
  - Local Institution - 0061, Las Palmas
  - Local Institution - 0074, Madrid
  - Local Institution - 0123, Madrid
  - Local Institution - 0042, Málaga
  - Local Institution - 0043, Valencia
- Switzerland (2):
  - Local Institution - 0015, Basel
  - Local Institution - 0104, Sankt Gallen
- United Kingdom (4):
  - Local Institution - 0135, Middlesbrough, Cleveland
  - Local Institution - 0101, London, Greater London
  - Local Institution - 0095, Manchester, Lancashire
  - Local Institution - 0067, Leicester

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04623775.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 468 Randomized and 463 Treated
Groups:
- Part 1: Treatment A: Nivo 360mg Q3W + Rela 720mg Q3W + Histology Based PDCT
- Part 1: Treatment B; Part 2: Treatment C: Nivo 360mg Q3W + Rela 360mg Q3W + Histology Based PDCT
- Part 2: Treatment D: Nivo 360mg Q3W + Histology Based PDCT
Period: Randomization
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 2: Treatment C | Part 2: Treatment D
Started | 79 | 80 | 158 | 151
Completed (Completed = Will Receive Treatment) | 77 | 79 | 158 | 149
Not Completed | 2 | 1 | 0 | 2
Not completed — No Longer Meets Study Criteria | 2 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 1
Not completed — Other Reasons | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 2: Treatment C | Part 2: Treatment D
Started | 77 | 79 | 158 | 149
Completed (= on going treatment) | 9 | 12 | 61 | 60
Not Completed | 68 | 67 | 97 | 89
Not completed — participant withdrew consent | 4 | 0 | 1 | 2
Not completed — Death | 3 | 1 | 4 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — poor/non compliance | 0 | 0 | 1 | 0
Not completed — participant no longer meets study criteria | 0 | 1 | 0 | 0
Not completed — administrative reasons by sponsor | 3 | 2 | 0 | 0
Not completed — other reasons | 2 | 0 | 1 | 1
Not completed — disease progression | 40 | 35 | 63 | 63
Not completed — study drug toxicity | 12 | 15 | 13 | 12
Not completed — AE unrelated to study drug | 4 | 9 | 12 | 9
Not completed — participant request to discontinue treatment | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Total
Number analyzed (Participants) | 79 | 80 | 158 | 151 | 468
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 42 | 73 | 72 | 224
  >=65 years | 42 | 38 | 85 | 79 | 244
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 55 | 57 | 172
  Male | 51 | 48 | 103 | 94 | 296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 12 | 31 | 28 | 87
  Not Hispanic or Latino | 37 | 44 | 91 | 88 | 260
  Unknown or Not Reported | 26 | 24 | 36 | 35 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 2 | 5
  White | 75 | 77 | 148 | 141 | 441
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 8 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: TRAEs Leading to Discontinuation Within 12 Weeks of First Dose in Part 1
Description: Percentage of participants with treatment related adverse events (TRAEs) leading to discontinuation within 12 weeks of first dose.
  AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: from first dose to 12 weeks after first dose
Population: All Treated Dose-Safety Evaluable participants in part 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 71 | 66
Percentage of Participants | 5.6 [1.6 to 13.8] | 12.1 [5.4 to 22.5]
Statistical Analysis 1: Comparison: Part 1: Treatment A vs Part 1: Treatment B; Test type: Superiority; Risk Difference (RD) = -6.5, 95% CI 2-sided [-16.0 to 3.0]

2. Primary Outcome: ORR Per RECISTS v1.1 by BICR in Part 2
Description: Objective Response Rate (ORR) per RECIST v1.1 by BICR is defined as the number of participants in the randomized population who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on BICR assessments (using RECIST v1.1) divided by the number of participants in the population. BOR is defined as the best response, as determined by the BICR, recorded between the date of randomization and the date of first objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first.
Time Frame: Approximately 14.8 Months
Population: All randomized participants in Part 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 151
Percentage of Participants | 50.6 [43.8 to 57.4] | 43.0 [36.2 to 50.1]
Statistical Analysis 1: Comparison: Part 2: Treatment C vs Part 2: Treatment D; Test type: Superiority; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.39, 90% CI 2-sided [0.94 to 2.05]

3. Secondary Outcome: TRAEs Leading to Discontinuation in Part 1
Description: Number of participants with treatment related adverse events (TRAEs) leading to discontinuation based on grade.
  AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be determined for severity according to the NCI CTCAE v5.0
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 32.8 Months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 77 | 79
Participants
  Any Grade | 21 | 18
  Grade 3 to 4 | 13 | 12
  Grade 5 | 1 | 0

4. Secondary Outcome: Number of Participants With a Treatment Related AEs in Part 1
Description: Number of participants with a treatment related AE in part 1.
  AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be determined for severity according to the NCI CTCAE v5.0
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 32.8 Months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 77 | 79
Participants | 75 | 76

5. Secondary Outcome: Number of Participants With Treatment Releted SAEs in Part 1
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose, results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [e.g., medical, surgical] to prevent one of the other serious outcomes listed in the definition).
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 32.8 Months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 77 | 79
Participants
  Any Grade | 20 | 24
  Grade 3 to 4 | 14 | 18
  Grade 5 | 2 | 4

6. Secondary Outcome: Number of Participants With Treatment Releted Select AEs in Part 1
Description: AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Select Adverse Events (AEs) will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 32.8 Months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 77 | 79
Participants
  Gastrointestinal | 18 | 15
  Hepatic | 26 | 18
  Pulmonary | 4 | 5
  Renal | 9 | 4
  Skin | 24 | 18
  Hypersensitivity/Infusion Reaction | 5 | 2

7. Secondary Outcome: ORR by PD-L1 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 2
Time Frame: Approximately 14.8 Months
Population: All randomized participants in Part 2
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 151
Percentage of Participants
  PD-L1 <1%: number analyzed (Participants) | 70 | 67
  PD-L1 <1% | 48.6 [38.2 to 59.0] | 44.8 [34.4 to 55.5]
  PD-L1 >= 1%: number analyzed (Participants) | 79 | 71
  PD-L1 >= 1% | 53.2 [43.3 to 62.8] | 39.4 [29.7 to 49.9]
  Not Quantifiable: number analyzed (Participants) | 9 | 13
  Not Quantifiable | 44.4 [16.9 to 74.9] | 53.8 [28.7 to 77.6]

8. Secondary Outcome: DoR Per RECISTS v1.1 by BICR in Part 2
Description: Duration of Response (DOR) will be assessed by BICR. It is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the first objectively documented tumor progression as determined by the BICR (per RECIST v1.1), or death due to any cause, whichever occurs first.
Time Frame: Approximately up to 13.7 months
Population: All randomized participants in Part 2
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 151
Months | 8.41 [7.43 to NA] — Upper limit was not reached due to an insufficient number of participants with events | 7.10 [5.62 to NA] — Upper limit was not reached due to an insufficient number of participants with events

9. Secondary Outcome: Number of Participants With a AE in Part 2
Description: Number of participants with an adverse event (AE).
  AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 14.8 Months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 149
Participants
  Any Grade | 158 | 147
  Grade 3 to 4 | 90 | 85
  Grade 5 | 26 | 19

10. Secondary Outcome: Number of Participants With a Treatment Related AEs in Part 2
Description: AE is defined as any new untoward medical occurrence or worsenig of a preexising medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 14.8 Months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 149
Participants
  Any Grade | 147 | 138
  Grade 3 to 4 | 79 | 78
  Grade 5 | 4 | 4

11. Secondary Outcome: Number of Participants With a Treatment Related SAEs in Part 2
Description: SAE is defined as a life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe). SAEs can also result in death. The AE requires inpatient hospitalization or causes prolongation of existing hospitalization. Results in persistent or significant disability/incapacity. Is a congenital anomaly/birth defect. Is an important medical event (defined as a medical event(s) that may not be immediately lifethreatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [e.g., medical, surgical] to prevent one of the other serious outcomes listed in the definition above.)
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 14.8 Months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 149
Participants
  Any Grade | 34 | 36
  Grade 3 to 4 | 26 | 28
  Grade 5 | 4 | 4

12. Secondary Outcome: Number of Participants With Endocrine Immune-mediated Adverse Events in Part 2
Description: IMAEs are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity.
  Grading will be determined for severity according to the NCI CTCAE v5.0.
Time Frame: From first dose to 30 days post last dose of study therapy (Approximately 14.8 Months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Treatment C | Part 2: Treatment D
Number analyzed (Participants) | 158 | 149
Participants
  Adrenal Insufficiency | 2 | 3
  Hypothyroidism/Thyroiditis | 22 | 13
  Hypothyroidism | 21 | 13
  Thyroiditis | 2 | 0
  Diabetes Mellitus | 1 | 0
  Hyperthyroidism | 14 | 3
  Hypophysitis | 0 | 1

13. Secondary Outcome: ORR by LAG-3 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 2
Time Frame: On Going
Reporting Status: Not Posted, anticipated posting 2027-01

14. Secondary Outcome: ORR by FG-L1 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 2
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

15. Secondary Outcome: PFS Per RECISTS v1.1 by BICR in Part 2
Description: Progression Free Survival is defined as the time between the date of randomization and the first date of documented progression, based on BICR assessments (per RECIST v1.1), or death due to any cause, whichever occurs first.
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

16. Secondary Outcome: PFS by PD-L1 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 15
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

17. Secondary Outcome: PFS by LAG-3 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 15
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

18. Secondary Outcome: PFS by FG-L1 Expression Per RECISTS v1.1 by BICR in Part 2
Description: as for outcome 15
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

19. Secondary Outcome: Number of Participants With Treatment Releted Select AEs in Part 2
Description: as for outcome 6
Time Frame: Ongoing
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: All-Cause mortality, Adverse Events and Serious Adverse Events: (From first dose to last dose + 135 days): Approximately 36 Months
Description: The number at Risk for All-Cause Mortality represents all Treated Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Part 1: Treatment A | Part 1: Treatment B | Part 2: Treatment C | Part 2: Treatment D
All-Cause Mortality (participants affected / at risk) | 47/77 | 46/79 | 79/158 | 70/149
Serious Adverse Events (participants affected / at risk) | 46/77 | 52/79 | 103/158 | 81/149
Other Adverse Events (participants affected / at risk) | 74/77 | 78/79 | 151/158 | 145/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Treatment A (N=77) | Part 1: Treatment B (N=79) | Part 2: Treatment C (N=158) | Part 2: Treatment D (N=149)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 6 | 3
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 10
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 4 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 3
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 3 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 3
Asthenia (General disorders) | 2 | 2 | 3 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 2 | 0 | 1 | 3
Disease progression (General disorders) | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 6 | 3 | 2
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 4 | 3
Sudden death (General disorders) | 1 | 0 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 3 | 0
Cholangitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 2 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 2 | 3 | 2
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 6 | 14 | 10
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Sepsis (Infections and infestations) | 3 | 2 | 0 | 4
Septic shock (Infections and infestations) | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Adenovirus test positive (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 1 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 | 40 | 36
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Treatment A (N=77) | Part 1: Treatment B (N=79) | Part 2: Treatment C (N=158) | Part 2: Treatment D (N=149)
Anaemia (Blood and lymphatic system disorders) | 51 | 43 | 109 | 92
Eosinophilia (Blood and lymphatic system disorders) | 4 | 0 | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 16 | 12
Leukopenia (Blood and lymphatic system disorders) | 11 | 12 | 17 | 16
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4 | 20 | 9
Neutropenia (Blood and lymphatic system disorders) | 28 | 29 | 38 | 38
Neutrophilia (Blood and lymphatic system disorders) | 2 | 0 | 10 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 16 | 47 | 34
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 9 | 1
Adrenal insufficiency (Endocrine disorders) | 2 | 5 | 3 | 3
Hyperthyroidism (Endocrine disorders) | 14 | 12 | 15 | 6
Hypothyroidism (Endocrine disorders) | 15 | 10 | 26 | 14
Lacrimation increased (Eye disorders) | 4 | 7 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 10 | 6 | 9 | 8
Constipation (Gastrointestinal disorders) | 29 | 17 | 33 | 20
Diarrhoea (Gastrointestinal disorders) | 26 | 18 | 34 | 30
Dry mouth (Gastrointestinal disorders) | 4 | 4 | 8 | 3
Dyspepsia (Gastrointestinal disorders) | 7 | 3 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 33 | 29 | 55 | 40
Stomatitis (Gastrointestinal disorders) | 6 | 4 | 4 | 4
Vomiting (Gastrointestinal disorders) | 17 | 16 | 27 | 20
Asthenia (General disorders) | 30 | 27 | 37 | 36
Chest pain (General disorders) | 5 | 3 | 7 | 5
Face oedema (General disorders) | 4 | 0 | 0 | 1
Fatigue (General disorders) | 33 | 25 | 43 | 37
General physical health deterioration (General disorders) | 3 | 4 | 2 | 5
Mucosal inflammation (General disorders) | 1 | 8 | 9 | 10
Non-cardiac chest pain (General disorders) | 7 | 1 | 5 | 8
Oedema peripheral (General disorders) | 11 | 8 | 17 | 18
Pain (General disorders) | 2 | 4 | 4 | 4
Peripheral swelling (General disorders) | 4 | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 11 | 18 | 11
Xerosis (General disorders) | 4 | 4 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 7 | 6 | 1 | 2
COVID-19 (Infections and infestations) | 10 | 6 | 4 | 4
Candida infection (Infections and infestations) | 3 | 4 | 1 | 3
Nasopharyngitis (Infections and infestations) | 5 | 0 | 4 | 1
Oral candidiasis (Infections and infestations) | 4 | 5 | 2 | 2
Pneumonia (Infections and infestations) | 5 | 3 | 8 | 5
Respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 2
Urinary tract infection (Infections and infestations) | 8 | 8 | 11 | 14
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 2 | 4 | 3
Alanine aminotransferase increased (Investigations) | 18 | 15 | 13 | 17
Aspartate aminotransferase increased (Investigations) | 16 | 15 | 14 | 17
Blood alkaline phosphatase increased (Investigations) | 7 | 7 | 10 | 4
Blood bilirubin increased (Investigations) | 5 | 6 | 4 | 2
Blood calcium increased (Investigations) | 5 | 6 | 0 | 1
Blood cholesterol increased (Investigations) | 4 | 2 | 7 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 5 | 7 | 8
Blood creatinine increased (Investigations) | 12 | 7 | 18 | 16
Blood glucose increased (Investigations) | 2 | 4 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 4 | 5 | 4 | 3
Blood magnesium decreased (Investigations) | 9 | 7 | 2 | 1
Blood potassium decreased (Investigations) | 4 | 4 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 5 | 4 | 6 | 1
Blood urea increased (Investigations) | 0 | 0 | 9 | 3
Gamma-glutamyltransferase increased (Investigations) | 5 | 3 | 11 | 3
Haemoglobin decreased (Investigations) | 5 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 4 | 5 | 1
Neutrophil count decreased (Investigations) | 17 | 10 | 19 | 12
Platelet count decreased (Investigations) | 19 | 13 | 22 | 17
Troponin T increased (Investigations) | 2 | 4 | 6 | 4
Troponin increased (Investigations) | 6 | 8 | 15 | 21
Weight decreased (Investigations) | 10 | 5 | 8 | 3
White blood cell count decreased (Investigations) | 6 | 3 | 12 | 5
Decreased appetite (Metabolism and nutrition disorders) | 21 | 24 | 27 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 4 | 19 | 8
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 8 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 6 | 8 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 4 | 7 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 7 | 8 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 7 | 16 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 11 | 12 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 5 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 11 | 26 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4 | 12 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 15 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 9 | 7
Dizziness (Nervous system disorders) | 5 | 7 | 13 | 11
Dysgeusia (Nervous system disorders) | 5 | 4 | 6 | 7
Headache (Nervous system disorders) | 13 | 11 | 12 | 13
Neuropathy peripheral (Nervous system disorders) | 5 | 7 | 15 | 7
Paraesthesia (Nervous system disorders) | 2 | 3 | 6 | 9
Anxiety (Psychiatric disorders) | 3 | 4 | 6 | 5
Insomnia (Psychiatric disorders) | 5 | 8 | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 19 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 18 | 15 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 8 | 12 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4 | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 7 | 8 | 16
Rash (Skin and subcutaneous tissue disorders) | 14 | 7 | 23 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 7 | 2 | 2
Hypertension (Vascular disorders) | 7 | 7 | 7 | 8
Hypotension (Vascular disorders) | 3 | 7 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04623775/Prot_SAP_001.pdf